CLINICAL TRIAL: NCT01491724
Title: The Learning Curve of Probe-based Confocal Laser Endomicroscopy (pCLE) Images Interpretation in Gastric Intestinal Metaplasia(GIM)
Brief Title: The Learning Curve of Probe-based Confocal Laser Endomicroscopy (pCLE) Images Interpretation in Gastric Intestinal Metaplasia (GIM)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principle investigator, King Chulalongkorn Memorial Hospital
Other Study IDs: RP001
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pCLE images

SUMMARY:
The Learning Curve of Probe-based Confocal Laser Endomicroscopy (pCLE) images interpretation in Gastric Intestinal Metaplasia (GIM)

Objective:

The aim of this study is to evaluate the learning curve of pCLE images interpretation in GIM.

Research design:

Blinded review of pCLE images for the diagnosis of GIM

Sample size:

Five beginner endoscopists will be assigned in this study to read approximately 80 videoclips

Data analysis:

ROC curve is analyzed by SPSS version 16.

Expected Benefit and Clinical Application Information on the learning curve for GIM interpretation from pCLE images in order to develop early gastric cancer detection

DETAILED DESCRIPTION:
Background and Rationale:

Gastric cancer remains the second leading cause of cancer related death in the world. The incidence and mortality rate is predominant in East Asia[1]. Usually, gastric cancer is asymptomatic in early stage; therefore, most patients are in the advanced stage and incurable at diagnosis. The pathogenesis of intestinal type gastric cancer is sequential and multistep pathway. Gastric intestinal metaplasia (GIM) is the precancerous lesion for intestinal type gastric cancer[2]. The strategies which can detect precancerous and/or early cancerous transformation are very beneficial because only early gastric cancer can potentially be cured by endoscopic treatment. Probe-based confocal laser endomicroscope or pCLE is useful for GIM detection with 94% in sensitivity[3]. However, this perfect sensitivity in pCLE interpretation is provided in only expertise. We still do not know how to be an expert in GIM interpretation. No study about learning curve in GIM interpretation by pCLE published

Observation and Measurement:

Collect the accuracy in GIM interpretation from pCLE reported in ROC curve

Methodology:

1. Six inexperienced pCLE readers were recruited.
2. All inexperienced pCLE readers must attend the learning session.
3. Self-review from CD is recommended for all inexperienced pCLE readers
4. Two-week interval for examination in GIM interpretation from 20 new histology-proved pCLE images (GIM and normal mucosa) for 5 sessions are on schedule after training session.
5. All Inexperienced pCLE readers need to review the training CD at least a day before each examination.
6. The accuracy rate in each examination will be recorded individually for each inexperienced pCLE reader.
7. ROC curve is reported for learning curve in GIM interpretation from pCLE images.

Data collection:

All data will be processed and recorded by one physician.

ELIGIBILITY:
Inclusion Criteria:

* First year fellow of gastroenterologist who never have the experienced in pCLE interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5 beginner endoscopists who never had the experience in pCLE
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The change of accuracy of pCLE images interpretation in GIM after each examination | Baseline and every 2 weeks for 4 sessions
  Percentage of accuracy changing in each examination

CONTACTS AND LOCATIONS:
Overall Officials: Rungsun Rerknimitr, Professor, Study Director — King Chulalongkorn Memorial Hospital; Rapat Pittayanon, MD, Principal Investigator — King Chulalongkron Memorial Hospital
Locations (1):
- Rapat Pittayanon, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: Related Info — http://www.medchulairb.com